CLINICAL TRIAL: NCT02901171
Title: The Contribution of a Smartphone Application to Acceptance and Commitment Therapy Group Treatment for Smoking Cessation: a Randomised Controlled Trial Investigating Its Efficacy, Mediators and Moderators
Brief Title: The Contribution of a Smartphone Application to Acceptance and Commitment Therapy Group Treatment for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: moconnor
Record Dates: First submitted 2016-09-09; First posted 2016-09-15 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Smoking
Keywords: Smoking cessation; Acceptance and Commitment Therapy; Smartphone
MeSH Terms: conditions — Smoking; Smoking Cessation

ARMS (3):
- Combined Treatment (Experimental): ACT group treatment combined with smartphone application
  Interventions: Behavioral: ACT group treatment combined with smartphone application
- Acceptance and Commitment Therapy (ACT) (Active Comparator): ACT group treatment
  Interventions: Behavioral: ACT group treatment
- Behavioural Support Programme (Active Comparator): Group based Behavioural Support Programme
  Interventions: Behavioral: Group based Behavioural Support Programme

INTERVENTIONS:
Behavioral: ACT group treatment combined with smartphone application — The Acceptance and Commitment Therapy (ACT) group treatment for smoking cessation will be delivered in six weekly 90-min sessions. Smoking cessation will be promoted in each session by targeting core processes of the ACT model including acceptance, cognitive defusion, mindfulness, flexible perspective taking, values clarification and committed action. In addition, participants will receive an ACT-based smartphone application for smoking cessation. The application will foster core processes of the ACT model through daily exercises, tips and tools.
  Arms: Combined Treatment
Behavioral: ACT group treatment
  Arms: Acceptance and Commitment Therapy (ACT)
Behavioral: Group based Behavioural Support Programme — The Behavioural Support Programme will be facilitated by stop smoking experts and delivered in six weekly 90-min sessions in a group format. During the sessions, advice, support and information on smoking cessation will be given to participants and behavioural techniques will be reviewed.
  Arms: Behavioural Support Programme

SUMMARY:
The purpose of this study is to evaluate the efficacy of a smartphone application in enhancing Acceptance and Commitment Therapy group treatment for smoking cessation. This study also aims to elucidate the processes through which the treatment promotes smoking cessation and for whom it is most effective.

DETAILED DESCRIPTION:
Smoking is the single biggest preventable cause of death in Ireland and costs the exchequer approximately €1-2 billion per annum. Currently, 19.2% of Irish people aged 15 and over smoke. Given the magnitude of human suffering and economic cost associated with smoking, the systematic empirical development of cost-effective smoking cessation interventions is a major public health need. Combining a group-based treatment for smoking cessation with a theoretically-consistent smartphone application has the advantage of augmenting therapeutic content delivered in the clinic with on-the-spot assistance in the individual's natural environment. In accordance, this study will evaluate the efficacy of a smartphone application in enhancing Acceptance and Commitment Therapy group treatment for smoking cessation. This study will also elucidate the processes through which the treatment promotes smoking cessation. Identifying such mediators of change can inform the enhancement of subsequent interventions, enabling them to retain efficacious elements and disregard redundant elements. Furthermore, this study will identify the participant characteristics associated with differential response to the treatment. Clarifying such treatment moderators can facilitate practitioners in selecting optimal treatments for individual service users.

Participants will attend a baseline assessment on an individual basis prior to their smoking cessation attempt. During this session, participants will provide a breath sample and complete a series of self-report measures: Fagerström Test of Nicotine Dependence, Commitment to Quitting Scale, smoking-related variables (e.g., years smoking, previous quit attempts, etc.), Avoidance and Inflexibility Scale, Mental Health Continuum-Short Form, Valuing Questionnaire, Present Moment Awareness Subscale of the Philadelphia Mindfulness Scale, and the Cognitive Fusion Questionnaire. Participants will then be randomly allocated to the combined treatment, ACT group treatment or group based Behavioural Support Programme. A post-treatment assessment will be conducted to investigate changes in the variables measured at baseline. In addition, a six-month follow-up assessment will determine whether the effects of the treatments are sustained over an extended period of time.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Interested in quitting smoking in the next 30 days
* Smoking 10 or more cigarettes per day for at least the past 12 months
* Daily access to a smartphone that is compatible with applications from iTunes (iPhone) or Google Play (Android)

Exclusion Criteria:

* Currently participating in another smoking cessation intervention
* Failure to the meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Seven-day point-prevalence abstinence | 6 weeks after beginning treatment
Seven-day point-prevalence abstinence | 6 months after beginning treatment

SECONDARY OUTCOMES:
Positive mental health measured by the Mental Health Continuum-Short Form | 6 weeks after beginning treatment
Positive mental health measured by the Mental Health Continuum-Short Form | 6 months after beginning treatment
Cigarettes per day in non-abstinent participants | 6 weeks after beginning treatment
Cigarettes per day in non-abstinent participants | 6 months after beginning treatment

CONTACTS AND LOCATIONS:
Overall Officials: Louise McHugh, Ph.D., Principal Investigator — University College Dublin
Locations (1):
- University College Dublin, Dublin, Leinster, Ireland

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700